CLINICAL TRIAL: NCT01790100
Title: A Randomized, Phase 2a, Partially-Blind, Dose-Ranging Study to Evaluate the Safety, Pharmacokinetics and Efficacy of VX-135 With Ribavirin in Treatment-Naïve Subjects With Chronic Hepatitis C
Brief Title: A Phase 2a, Dose-Ranging Study to Evaluate the Safety, Pharmacokinetics and Efficacy of VX-135 With Ribavirin in Treatment-Naïve Subjects With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALS-135-101; 2012-005633-37 (EudraCT Number)
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- VX-135 low dose in combination with ribavirin (Experimental): 12 weeks of VX-135 in combination with ribavirin
  Interventions: Drug: VX-135; Drug: Ribavirin
- VX-135 high dose in combination with ribavirin (Experimental)
  Interventions: Drug: VX-135; Drug: Ribavirin

INTERVENTIONS:
Drug: VX-135 — 12 weeks of VX-135
Drug: Ribavirin — 12 weeks of ribavirin

SUMMARY:
The purpose of the study is to determine the safety, pharmacokinetics and efficacy of orally administered VX-135 with ribavirin in treatment naive subjects with chronic hepatitis C infection.

DETAILED DESCRIPTION:
Up to twenty (20) subjects with CHC GT1 infection will be randomized in a 1:1 ratio (with stratification by IL-28B genotype (CC versus non-CC)) to evaluate VX-135 low dose or high dose both given in combination with RBV for 12 weeks.

Safety and tolerability will be evaluated on an ongoing basis through assessment of adverse events (AEs), lab evaluations and physical examinations. Subjects will be monitored from Day 1 through end of follow-up for virologic breakthrough or relapse.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects (male and female) must be between 18-60 years of age
* Subjects must have Chronic Hepatitis C
* Subjects must be treatment naive
* Subjects must have laboratory values at screening within limits as specified by the protocol

Key Exclusion Criteria:

* Evidence of cirrhosis
* Female subjects who are pregnant or nursing or male subjects with a female partner of childbearing potential who is unwilling to adhere to the contraception requirements, is pregnant or nursing, or planning to become pregnant during the study
* any other cause of significant liver disease in addition to hepatitis C
* Diagnosis of or suspected hepatocellular carcinoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Safety | Week 12
  The safety and tolerability as assessed by evaluating adverse events and laboratory testing.

SECONDARY OUTCOMES:
evidence of HCV RNA viral load reduction | 16 weeks
  The proportion of subjects who have an SVR at 4 weeks after the last planned dose of treatment (SVR4)

CONTACTS AND LOCATIONS:
Locations (1):
- Arensia, Republican Clinical Hospital, Chisinau, Moldova